CLINICAL TRIAL: NCT06162936
Title: Neutrophil Oxidative Burst in Early and Late Onset Pediatric Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute for Mother and Child Health Alessandrescu Rusescu (Other)
Collaborators: Marie Curie Emergency Children's Hospital, Bucharest (Unknown); Victor Gomoiu Children's Hospital, Bucharest (Unknown)
Responsible Party: Sponsor
Other Study IDs: IBD20232024
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Chronic Granulomatous Disease
Keywords: inflammatory bowel disease; chronic granulomatous disease; inborn errors of immunity
MeSH Terms: conditions — Granulomatous Disease, Chronic; Inflammatory Bowel Diseases | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inflammatory bowel disease patients: Pediatric patients (under 18 years of age) diagnosed with IBD
  Interventions: Diagnostic Test: Phagoburst; Diagnostic Test: Lymphocytes subsets; Diagnostic Test: Genetic testing
- Healthy controls: Healthy chidren (no chronic disease)
  Interventions: Diagnostic Test: Phagoburst

INTERVENTIONS:
Diagnostic Test: Phagoburst — The main objective is to perform oxidative burst activity in pediatric patients with a definitive diagnosis of IBD and compare them with healthy controls.
Diagnostic Test: Lymphocytes subsets — To determine lymphocytes subsets in patients with suspicion of IEI
  Groups: Inflammatory bowel disease patients
Diagnostic Test: Genetic testing — Perform targeted genetic testing in those with reduced to absent oxidative activity in search of PIDs and susceptibility variants
  Groups: Inflammatory bowel disease patients

SUMMARY:
ABSTRACT Introduction Residual or absent oxidase function in peripheral neutrophils may point to an inborn defect of neutrophil function - chronic granulomatous disease (CGD) - whereas low to normal oxidative burst capacity has been linked to variants in various members of the NADPH-complex.

Aims To assess the clinical value of routinely measuring oxidative burst activity of granulocytes in pediatric patients diagnosed with very early onset IBD (VEO-IBD) and late onset IBD.

Objectives To investigate possible correlations between neutrophil function and IBD disease activity and to inquire the presence of genetic variants in those with low to absent oxidative burst. To identify the rate of monogenic VEO-IBD in our cohort.

Materials and Methods The proposal constitutes a collaborative effort among Romanian pediatric tertiary care centers to examine the value of assessing neutrophil function in all pediatric IBD patients. Children aged <18 years diagnosed with Crohn's disease, ulcerative colitis or IBD-undetermined and age-matched healthy controls are recruited. A DHR flow cytometry assay is performed in included subjects and controls. Reduced or absent burst activity will lead to genetic testing in search of overt immunodeficiency or susceptibility variants. All VEO-IBD patients will have an immunological work-up in search of a primary immunodeficiency.

Expected Results We anticipate to include a number of 150 pediatric patients with IBD over 12 months from the three pediatric gastroenterology units in Bucharest, Romania. We expect to identify an overall diminished neutrophil function in IBD patients versus controls and possible variants in the NADPH-complex genes.

ELIGIBILITY:
Inclusion Criteria:

Subjects:

1. age under 18 years;
2. confirmed diagnosis of IBD fulfilling standard diagnosis criteria (clinical, radiological, endoscopical, histological features)
3. parental/guardian consent for study enrollment

Controls:

Healthy age-gender matched controls

Exclusion Criteria:

1. IBD associated to an already defined monogenic defect
2. Diagnosis of IBD uncertain
3. HIV/TB positive

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will include pediatric patients diagnosed with IBD (right from the diagnosis or anytime during the disease course) from three different gastroenterology units in Bucharest, Romania.
  Screening tests for an imunological disease (neutrophil oxidative burst, lymphocyte subsets) will be performed in included patients and healthy controls by the home institution.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Oxidative burst activity in IBD patients | 12 months
  Perform oxidative burst activity in pediatric patients with a definitive diagnosis of IBD and compare them with healthy controls.
Genetic testing in patients with suspicion of IEI | 12 months
  Perform targeted genetic testing in those with reduced to absent oxidative activity in search of PIDs and susceptibility variants

SECONDARY OUTCOMES:
Role of burst activity in disease phenotype | 12 months
  Find correlations between burst activity and disease activity

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute for Mother and Child Health Alessandrescu Rusescu, Bucharest, County, Romania